CLINICAL TRIAL: NCT07246616
Title: Efficacy and Safety of CO₂ Laser Therapy Combined With Collagen Cream in Managing Vulvo-Vaginal Atrophy: A Randomized, Controlled Study on Symptom Relief and Microbiome Modulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Social Security, Republic of San Marino (Other)
Responsible Party: Principal Investigator, MAURIZIO FILIPPINI, Dott. Maurizio Filippini, Institute for Social Security, Republic of San Marino
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MF-01-24 1; N/1 (Other: UOC di Ostetricia e Ginecologia, Ospedale di Stato della Repubblica di San Marino, Istituto per la Sicurezza Sociale (I)
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Vulva; Atrophy
Keywords: Vulva; Atrophy; Co2; Vulvo-vaginal; Microbiome; Modulation; Laser; Theraphy; Collagen; Collagen Cream
MeSH Terms: conditions — Atrophy | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This is an interventional, single-center study. Patients will be randomized into two groups: one called the "control" group, in which patients will receive only the SmartXide2 treatment, and the second called "PALINGEN," in which patients will receive SmartXide2 treatment plus the application of Palingen cream. It should be noted that both SmartXide2 and Palingen cream (and their combination) have been part of the standard clinical practice at the experimental center for several years.
  The effectiveness of the combined action of the two treatments will be evaluated by analyzing the associated symptoms using a Visual Analogue Scale (VAS) from 1 to 10 for each symptom, as well as through analysis of the vaginal microbiome. Additionally, all adverse events will be recorded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laser Therapy Only (Control Group) (Active Comparator): Participants receive fractional CO₂ laser therapy according to the standard protocol for vulvo-vaginal atrophy.
  No additional topical treatment is applied.
  Laser sessions are performed at baseline (Day 0), Day 30, and Day 60.
  Follow-up visits include clinical evaluation and microbiome sampling at each time point.
  Interventions: Device: SmartXide2 treatment plus the application of Palingen cream; Device: Laser Therapy Only (Control Group)

INTERVENTIONS:
Device: SmartXide2 treatment plus the application of Palingen cream — Patients will be randomized into two groups: one called the "control" group, in which patients will receive only the SmartXide2 treatment, and the second called "PALINGEN," in which patients will receive SmartXide2 treatment plus the application of Palingen cream.
Device: Laser Therapy Only (Control Group) — Participants receive fractional CO₂ laser therapy according to the standard protocol for vulvo-vaginal atrophy.
  No additional topical treatment is applied.
  Laser sessions are performed at baseline (Day 0), Day 30, and Day 60.
  Follow-up visits include clinical evaluation and microbiome sampling at each time point.

SUMMARY:
This study evaluated a new treatment for postmenopausal women suffering from vulvo-vaginal atrophy (VVA), a condition that causes dryness, burning, and pain. Researchers tested whether combining CO₂ laser therapy with a collagen-based cream could improve symptoms more effectively than laser treatment alone.

DETAILED DESCRIPTION:
Sixty women participated in the study. Results showed that the combination treatment provided greater relief from discomfort and helped restore vaginal health, with fewer side effects. This approach may offer a safe and effective alternative for women who cannot use hormone-based therapies.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with absence of menstrual cycle for at least 12 months, diagnosed with vulvovaginal atrophy (VVA) and presenting with related symptoms such as dryness, introital and deep dyspareunia, bleeding during intercourse, itching, or burning related to the severity of VVA, whether spontaneous or drug-induced (radio- or chemotherapy), either with a single symptom or a combination thereof.
* Age between 35 and 75 years;
* Patients unresponsive or dissatisfied with previous topical estrogen therapy, or presenting contraindications to the use of local and/or systemic estrogens.
* Previous negative Pap test performed within 3 years prior to study enrollment.

Exclusion Criteria:

* • Pregnancy or breastfeeding;

  * Presence of preneoplastic or neoplastic lesions of the cervix, vagina, or vulva;
  * Presence of active genital and/or urinary tract infection;
  * Relative or absolute dermatological contraindications to laser use;
  * Ongoing hormonal therapy (systemic or local);
  * Neurological and/or psychiatric disorders;
  * Chronic systemic autoimmune or metabolic diseases;
  * Refusal to provide informed consent.

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Improvement in VVA (Vulvo-Vaginal Atrophy) symptoms | Outcome: Improvement in symptoms associated with vulvo-vaginal atrophy (VVA) Assessment Tool: Visual Analogue Scale (VAS) Time Frame: Baseline (Day 0) - before treatment Visit 1 (Day 30) - after first month of treatment Visit 2 (Day 60) - after second
  Assessed after 30 and 60 days of treatment using the Visual Analogue Scale (VAS).
  The VAS was used to quantify symptom intensity such as burning, dryness, itching, dyspareunia, and pain.
  Improvement was measured as the difference in VAS scores before and after treatment.

SECONDARY OUTCOMES:
Vaginal Microbiome Composition | Baseline (Day 0) - before treatment Visit 1 (Day 30) - after first month of treatment Visit 2 (Day 60) - after second month / end of treatment
  Analysis before and after 30 and 60 days of treatment.
  Parameters included:
  Biodiversity (Observed Operational Taxonomic Units, OTUs).
  Relative abundance of Lactobacillus genus and its species (L. crispatus, L. iners, etc.).
  Relative amounts of pathogenic bacteria (Gardnerella vaginalis, Atopobium vaginae, etc.).
Symptom improvement at intermediate time points | Baseline → Visit 1 (Day 30) Baseline → Visit 2 (Day 60)
  Comparison of VAS scores at Visit 1 (30 days) and Visit 2 (60 days) against baseline.
Adverse Events Monitoring | Continuous from first laser session (Day 0) through 30 days and 60 days post-treatment
  Frequency and severity of side effects (e.g., redness, mild bleeding, burning, swelling) were recorded throughout the study.

CONTACTS AND LOCATIONS:
Locations (1):
- UOC di Ostetricia e Ginecologia, Ospedale di Stato della Repubblica di San Marino, Istituto per la Sicurezza Sociale (ISS), San Marino, Borgo Maggiore, San Marino

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mueck AO, Ruan X, Prasauskas V, Grob P, Ortmann O. Treatment of vaginal atrophy with estriol and lactobacilli combination: a clinical review. Climacteric. 2018 Apr;21(2):140-147. doi: 10.1080/13697137.2017.1421923. Epub 2018 Jan 30. PMID 29381086
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29381086/